CLINICAL TRIAL: NCT04485806
Title: The Effect of Culture Media Microdroplet Geometry and Different Oil Overlay on Pre Implantation Embryonic Development in Dry Incubators: Prospective Randomized Study.
Brief Title: Culture Media Microdroplet Geometry With Different Oil Overlay and Its Effect on Embryonic Development.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MH0002
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Embryonic Development; Infertility
Keywords: dry incubator; Osmolality; Oil overlay; Microdrops
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Effect of two different culture dishes with two different oil overlay which used in human embryos culturing through ICSI procedures on the pre implantaion embryonic development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GPS / LM versus SPL/LM (Other): to determine the effect of micro droplet geometry in 3D dishes (GPS) or 2D dishes (SPL) in combination with light mineral oil (LM).
  Interventions: Other: GPS/LM; Other: SPL/LM
- GPS/PO versus SPL/PO (Other): to determine the effect of micro droplet geometry in 3D dishes (GPS) or 2D dishes (SPL) in combination with paraffin oil (PO).
  Interventions: Other: GPS/PO; Other: SPL/PO
- GPS/PO versus GPS/LM (Other): to determine the effect of oil overlay light mineral(LM) or paraffin oil (PO) in combination with paraffin oil 3D dishes (GPS).
  Interventions: Other: GPS/LM; Other: GPS/PO
- SPL/PO versus SPL/LM (Other): to determine the effect of oil overlay light mineral(LM) or paraffin oil (PO) in combination with paraffin oil 2D dishes (SPL).
  Interventions: Other: SPL/LM; Other: SPL/PO

INTERVENTIONS:
Other: GPS/LM — Media microdroplet geometry (3D dishes) in combination with light mineral oil overlay
  Arms: GPS / LM versus SPL/LM; GPS/PO versus GPS/LM
Other: SPL/LM — Media microdroplet geometry (2D dishes) in combination with light mineral oil overlay
  Arms: GPS / LM versus SPL/LM; SPL/PO versus SPL/LM
Other: GPS/PO — Media microdroplet geometry (3D dishes) in combination with Paraffin oil overlay
  Arms: GPS/PO versus GPS/LM; GPS/PO versus SPL/PO
Other: SPL/PO — Media microdroplet geometry (2D dishes) in combination with paraffin oil overlay
  Arms: GPS/PO versus SPL/PO; SPL/PO versus SPL/LM

SUMMARY:
A prospective randomized study included 1695 MII sibling oocytes collected from 100 patients undergoing ICSI.

DETAILED DESCRIPTION:
Purpose:

to determine the effect of culture media microdroplet geometry of different culture dishes and oil overlay on the pre implantation embryo development in dry incubators

Method:

We used sibling oocytes splits between two different dishes : GPS (life global, USA) and SPL (life science, Korea) with two different oils : light mineral oil (LM)(Irvine, USA) and paraffin oil (PO)(Vitro life, Sweden). All embryos cultured in dry incubators at the same conditions.

statistical analysis done using SPSS version 23

ELIGIBILITY:
Inclusion Criteria:

* Female age is ≤ 37 years old with ≥ 8 MII oocytes
* Males with normal semen parameters (WHO 2010).
* We conducted three experiments all with Siblings oocytes splits and all embryos

Exclusion Criteria:

* Oocyte or sperm donation.
* Sever male factor.
* Any contradictions to undergoing in vitro fertilization or goandotropin stimulation.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Blastulation rate | 5-6 days after ICSI
  Percentage of total blastocysts / Total cleaved embryos
High quality blast rate | 5-6 days after ICSI
  Morphological grading of trophectoderm and Inner cell mass using Gardner's criteria 1999, from grade A and B ( A is the highest quality). Total high grade embryos/ total blast embryos.

SECONDARY OUTCOMES:
Fertilization rate | 16-19 hours of ICSI
  Percentage of fertilized oocyte (appearance of two pronuclei) / Number of injected oocytes
Cleavage rate | 72 hours of ICSI
  Percentage of cleaved embryos/ total number of fertilized oocytes
High quality D3 embryos | 72 hours of ICSI
  High quality D3 embryos according to Gardner's criteria / total cleaved embryos
Good quality trophectoderm/inner cell mass | 5-6 days after ICSI
  better grade than 3BB of blast embryos according to Gardner's criteria 1999

CONTACTS AND LOCATIONS:
Overall Officials: Manar M Hozyen, MSc., Principal Investigator — Ganin Fertility Center; Amr Elshimy, BSc., Principal Investigator — Ganin Fertility Center; Hanaa Elkhader, BSc., Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc., Study Chair — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Egypt